CLINICAL TRIAL: NCT06401590
Title: Sensitivity and Predictive Value of Frozen Section of Sentinel Lymph Node Biopsy in Post Neoadjuvant Setting
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Fatima Safdar, PRINCIPAL INVESTIGATOR, Aga Khan University
Other Study IDs: 2022-7303-20844
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Lymph Node Metastasis; Breast Cancer
MeSH Terms: conditions — Lymphatic Metastasis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POSITIVE CASES
  Interventions: Diagnostic Test: FROZEN SENTINEL LYMPH NODE BIOPSY
- NEGATIVE CASES
  Interventions: Diagnostic Test: FROZEN SENTINEL LYMPH NODE BIOPSY

INTERVENTIONS:
Diagnostic Test: FROZEN SENTINEL LYMPH NODE BIOPSY — FROZEN SENTINEL LYMPH NODE BIOPSY

SUMMARY:
Axillary lymph node status is one of the most important prognostic factors in primary breast carcinomas. Sentinel lymph node biopsy has been increasing in post neoadjuvant setting when axillary nodes show good clinical and radiological response. It allows to determine the axillary lymph node status, which if negative, saves the patient from axillary dissection (AD) and its potential complications. To assess tumor response to neoadjuvant chemotherapy in the SLN, pathological evaluation is the gold standard. Response to neoadjuvant systemic therapy is an excellent predictor of outcome, and achievement of pathological complete response (PCR) in the SLN is a prognostic predictor of long-term outcome with significantly better disease-free survival and overall survival. Post-treatment isolated tumor cells (ITCs) and micro metastases predict worse survival compared with the same findings in the non-neoadjuvant setting. Histologically partial response to therapy, is characterized by small clusters and individual tumor cells set in hyaline stromal fibrosis. Most false negative cases had metastatic foci identified exclusively on permanent sections and are not due to a true diagnostic interpretation error. The timing of further axillary surgery, immediate or a subsequent operation should be routinely discussed at centers using intraoperative assessment of the sentinel lymph nodes, along with the potential for negative intraoperative findings and positive nodes on final pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients greater than 18 years of age
2. All diagnosed breast carcinoma patients ranging from T1 to T4 and N0 to N1, who have received neoadjuvant chemotherapy will be included.

Exclusion Criteria:

1. Poorly preserved biopsy material, insufficient to assess all the histological features.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were initially diagnosed with breast cancer greater than 18 years, stage T1 to T4, N0 to N1 by Section of Histopathology, Aga Khan University Hospital, Karachi from 2021 to 2022 and subsequently received neoadjuvant chemotherapy, were included.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with discrepant frozen and permanent biopsy results | From frozen section report to permanent section biopsy report, upto 1 week.
  The results of patient's frozen biopsy report and permanent section biopsy report will be compared and sensitivity, predictive value and false negative rate of frozen section biopsy will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ROMANA IDRESS, MBBS, FCPS, Principal Investigator — AKU
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Demographic details including age, diagnosis and results including sensitivity, specificity, and false negative rate of frozen SLNB after neoadjuvant chemotherapy.